CLINICAL TRIAL: NCT04339192
Title: Minimally Invasive Tricuspid Surgery Versus Medical Treatment for Severe Tricuspid Regurgitation After Left-sided Valve Surgery
Brief Title: Minimally Invasive Tricuspid Surgery vs Medical Treatment for Severe TR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2020-036R
Record Dates: First submitted 2020-04-05; First posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery group (Experimental): receiving minimally invasive tricuspid surgery including tricuspid valve replacement or repair plus medical treatment.
  Interventions: Procedure: Minimally Invasive Tricuspid Surgery
- Medical group (No Intervention): receiving medical treatment only

INTERVENTIONS:
Procedure: Minimally Invasive Tricuspid Surgery — minimally invasive tricuspid surgery including endoscopy-assist right minithoracotomy, vacuum-assist single femoral venous drainage without dissecting or snaring vena cava, direct right atriotomy through pericardium and the beating-heart technique.
  Arms: Surgery group

SUMMARY:
Late tricuspid regurgitation (TR) is a common complication after left-sided valve surgery (LSVS), which usually progresses slowly and results in right heart failure at terminal stage. Over the past 3 decades, with the advances in minimally invasive surgical techniques, operative mortality after reoperation for severe TR has significantly decreased from 30% to 3-8%, leading to a gradual shift from medical therapy alone to surgery in those patients. However, there has been no consensus on the clinical benefit of minimally invasive tricuspid surgery over medical therapy for severe TR after LSVS.

DETAILED DESCRIPTION:
In this multi-center randomized controlled trial, patients with severe TR after LSVS will be recruited. The patients will be randomly assigned to surgery plus medical therapy (surgery group) or medical therapy alone (control group). The primary outcome will be a composite of all-cause mortality, re-admission for right heart failure or the composite. Furthermore, echocardiography-based measurement of right heart function, New York Heart Association functional class, liver and kidney function, and quality of life will be compared between the 2 groups. All outcomes will be assessed at baseline and 6, 12 and 24 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Severe tricuspid regurgitation, as assessed by the clinical site echocardiographer using the transthoracic echocardiography.
2. A history of LSVS, including one or multiple procedures of aortic and/or mitral valve repair and/or replacement.
3. Left ventricular ejection fraction (LVEF) >45%, systolic pulmonary artery pressure <60 mmHg with pulmonary vascular resistance <6 woods unit.
4. Age ≥ 18 years.
5. Able to sign Informed Consent forms.

Exclusion Criteria:

1. TR due to: infective endocarditis, congenital tricuspid valve malformation, secondary to correction of congenital heart disease.
2. Left-sided valve dysfunction or coronary artery disease requiring concomitant procedures.
3. Prior surgical or percutaneous tricuspid valve intervention.
4. Evidence of an acute myocardial infarction in the prior 90 days
5. Contraindications to cardiopulmonary bypass or the expected operative mortality >30% (calculated by the Society of Thoracic Surgeons score or the EuroSCORE II).
6. Any comorbidity with life expectancy <2 years
7. Recent history of psychiatric disease (including drug or alcohol abuse) that is likely to impair compliance with the study protocol.
8. Pregnancy at the time of randomization.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
the rate of all-cause death, re-hospitalization due to right heart failure or both of them | 2 years
  the rate of all-cause death, re-hospitalization due to right heart failure or both of them

SECONDARY OUTCOMES:
right heart function | 2 years
  echocardiography-based measurement of right heart function
New York Heart Association functional class | 2 years
  New York Heart Association functional class including I, II, III, IV class
liver function | 2 years
  total bilirubin, conjugated bilirubin
liver function | 2 years
  prealbumin.
kidney function | 2 years
  blood urea nitrogen
kidney function | 2 years
  creatinine
kidney function | 2 years
  uric acid.
life quality scores | 2 years
  quality of life using the SF-12 form

CONTACTS AND LOCATIONS:
Overall Officials: Chunsheng Wang, MD, Principal Investigator — Zhongshan Hospital, Fudan Univerisity
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Now we have decided not to make IPD available to other researchers.

REFERENCES:
- [Background] Chen J, Hu K, Ma W, Lv M, Shi Y, Liu J, Wei L, Lin Y, Hong T, Wang C. Isolated reoperation for tricuspid regurgitation after left-sided valve surgery: technique evolution. Eur J Cardiothorac Surg. 2020 Jan 1;57(1):142-150. doi: 10.1093/ejcts/ezz160. PMID 31157373